CLINICAL TRIAL: NCT03563911
Title: Brief Mindfulness-Based Intervention for Chronic Pain: A Pilot Randomized Clinical Trial
Brief Title: Brief Mindfulness and Nutrition-Based Interventions for Chronic Pain: Strategies to Ease Pain
Acronym: STEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0864; A532007 (Other: UW Madison); SMPH/FAMILY MED/RES GRANTS (Other: UW Madison); Protocol Version 6/25/2018 (Other: UW Madison)
Record Dates: First submitted 2018-05-07; First posted 2018-06-20 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Opioid Use; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Mindfulness-Based Intervention (Experimental): Those assigned to the Brief Mindfulness-Based Intervention (BMBI) Arm will receive BMBI.
  Interventions: Behavioral: Brief Mindfulness-Based Intervention (BMBI)
- Control/Nutrition Education (Active Comparator): Those assigned to the Control/Nutrition Education Arm will receive the nutrition education intervention.
  Interventions: Behavioral: Control/Nutrition Education

INTERVENTIONS:
Behavioral: Brief Mindfulness-Based Intervention (BMBI) — The BMBI is be based on a BMBI which demonstrated analgesic effects in a previous study. Relative to full-length interventions, we will employ a brief intervention; the 20-minute BMBI session will include education on the foundational concepts of mindfulness and its relevance to chronic pain (5 minutes) and a guided mindfulness practice involving focused attention on the breath and monitoring of thoughts, feelings, and body sensations (15 minutes). BMBI participants will be encouraged to practice the taught mindfulness technique at home at least 20 minutes/day for 1 week (a handout and link to an online guided mindfulness practice will be provided).
  Arms: Brief Mindfulness-Based Intervention
Behavioral: Control/Nutrition Education — The Control intervention will involve nutrition education, adapted from an existing manual of cognitive-behavioral therapy for opioid-treated chronic pain. Control intervention protocol will match the BMBI in terms of time / structure to control for the non-specific, non-mindfulness effects of BMBI. The 20-minute Control session will include education on the relationship between diet and pain (10 minutes) and recommendations for a healthy diet (10 minutes). Control participants will be encouraged to prepare healthy meals at home at least 20 minutes/day for 1 week (a handout and link to online resources will be provided).
  Arms: Control/Nutrition Education

SUMMARY:
This pilot randomized clinical trial (RCT) will randomize adults with chronic pain to one, 20-minute session of either: Brief Mindfulness-Based Intervention (BMBI) mindfulness training or nutrition education (Control). Following the session, participants will be encouraged to practice a technique associated with their intervention (i.e., practicing mindfulness technique in BMBI, preparing healthy meals in Control) 20 minutes/day for one week at home. Quantitative sensory testing (with cold pressor and algometer) will be conducted before and after the session, and self-reported outcome assessments will be conducted before and after the session and at 1-week follow-up.

DETAILED DESCRIPTION:
Participants. To gather pilot data on the effects of BMBI, the investigators will aim to enroll up to 60 participants (up to 30 in each condition). Participants will be adults with chronic non-cancer pain (daily pain for at least 3 months).

Outcomes. Outcome measures were selected based on existing recommendations, including IMMPACT guidelines, for efficacy trials in chronic pain.

* Aim #1: Test the effects of BMBI, relative to control, on central pain processing using quantitative sensory testing. Quantitative sensory testing (cold pressor test and pressure algometer) will be used to characterize pain processing: pain threshold (i.e., when pain is first detected), pain tolerance (i.e., the duration of time that pain can be tolerated), and pain severity (i.e., intensity of pain). In the cold pressor test, a participant will be asked to place his or her hand in an ice bath until the pain is too great to remain in the water. Consistent with past research, a 15 liter refrigerated circulator (Polyscience MX15R-30-A11B) with water temperature set as low as 1°C will be used. In the pressure algometer test, the algometer will be used to apply pressure to the skin until the pain can no longer be tolerated. The investigators will utilize a device widely used in alogmeter pain research (Wagnder Force One Alogmeter FIPX).
* Aim #2: Test the immediate effects of BMBI, relative to control, on state self-report measures of pain, negative affect, and decentering. State self-report outcomes include: state decentering (7-item Decentering Subscale of the Toronto Mindfulness Scale), state pain intensity (1 item from the Brief Pain Inventory), state pain unpleasantness (1-item rated on 0-10 scale), state anxiety (1-item rated on 0-10 scale), state distress (1-item rated on 0-10 scale), state relaxation (1-item rated on 0-10 scale), and outcome expectancies (5-item Outcome Expectancies Questionnaire).
* Aim #3: Test longer-term effects of BMBI, relative to control, on trait self-report measures of pain, negative affect, trait mindfulness, and well-being. Trait self-report outcomes include: pain intensity and interference (9-item Brief Pain Inventory), anxiety and depression (14-item Hospital Anxiety and Depression Scale), trait mindfulness (15-item Mindful Attention Awareness Scale), psychological well-being (10-item Schwartz Outcome Scale), and home practice over the 4-week follow-up period (TLFB method).

Procedure. Participants will be recruited primarily via flyers and postings in newspapers and on the Internet. Prospective participants will be screened by phone (about 30 minutes). Provisionally eligible participants will be asked to attend a 1-hour appointment, which will begin with informed consent procedures (5-10 minutes) and a pre-intervention assessment (about 20 minutes; includes demographics questionnaire, self-report outcome measures, and quantitative sensory testing).

Eligible participants will be randomized to a condition, complete a 20-minute session of either BMBI or Control, and undergo a postintervention assessment (about 10 minutes; includes self-report outcome measures and quantitative sensory testing). Following the assessment, participants will be encouraged to practice the technique associated with their intervention (i.e., practicing mindfulness technique in BMBI, preparing healthy meals in Control) 20 minutes/day for 1 week at home and to track their practice and opioid use during the follow-up period; the follow-up assessments will be conducted over the phone by a research assistant and include the self-report outcome measures (no quantitative sensory testing). All study procedures are anticipated to last 2 hours and 30 minutes (30 minutes for screening, 1 hour for in-person appointment, and 30 minutes for each follow-up assessment).

Interventions: The BMBI is be based on a BMBI which demonstrated analgesic effects in a previous study. Relative to full-length interventions, the investigators will employ a brief intervention (i.e., one, 20-minute session) that could be delivered in routine clinical care, e.g., in primary care, and that could overcome cost and time/effort barriers associated with longer treatments. The 20-minute BMBI session will include education on the foundational concepts of mindfulness and its relevance to chronic pain (5 minutes) and a guided mindfulness practice involving focused attention on the breath and monitoring of thoughts, feelings, and body sensations (15 minutes). BMBI participants will be encouraged to practice the taught mindfulness technique at home at least 20 minutes/day for 1 week (a handout and link to an online guided mindfulness practice will be provided).

The Control intervention will involve nutrition education, adapted from an existing manual of cognitive-behavioral therapy for opioid-treated chronic pain. Control intervention protocol will match the BMBI in terms of time / structure to control for the non-specific, non-mindfulness effects of BMBI. The 20-minute Control session will include education on the relationship between diet and pain (10 minutes) and recommendations for a healthy diet (10 minutes). Control participants will be encouraged to prepare healthy meals at home at least 20 minutes/day for 1 week (a handout and link to online resources will be provided).

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. ≥ 18 years old
3. Chronic non-cancer pain (daily pain for at least 3 months)
4. Average daily pain score ≥3 on a 0-10 numerical rating scale (question from the Brief Pain Inventory)
5. Treatment with ≥30 mg/day of morphine-equivalent dose for ≥3 months
6. Capable of giving informed consent
7. Willing to complete all study activities

Exclusion Criteria:

1. Cancer pain
2. Current pregnancy
3. Diagnosed with psychotic or bipolar (mania) disorders ("active" in the prior 12 months)
4. Inability to safely or reliably participate in the study
5. Regular mindfulness meditation practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Cold pressor testing | 1 hour
  Cold pressor testing will be used to characterize pain processing (e.g., pain threshold, pain tolerance, pain severity). In the cold pressor test, a participant is asked to place his or her hand and forearm in an ice bath until the pain is too great to remain in the water. Consistent with past research, a 15 liter refrigerated circulator (Polyscience MX15R-30-A11B) with water temperature set as low as 1°C will be used in the present study.
Pressure algometer testing | 1 hour
  Pressure algometer testing will be used to characterize pain processing (e.g., pain threshold, pain tolerance, pain severity). In the pressure algometer test, the algometer is used to apply pressure to the skin until the pain can no longer be tolerated. In the current study, we will utilize a device widely used in alogmeter pain research (Wagnder Force One Alogmeter FIPX).
Brief Pain Inventory | 4 weeks
  Measures: 1) pain severity= mean of items 3-6 (ranges from 0-10 with higher scores indicating greater pain severity), and 2) pain interference= mean of items 9A-9G (ranges from 0-10 with higher scores indicating greater pain interference).
Hospital Anxiety and Depression Scale | 4 weeks
  Measures: 1) Anxiety (sum of 7 items; ranges from 0-21, with higher scores indicating greater anxiety), and 2) Depression (sum of 7 items; ranges from 0-21, with higher scores indicating greater depressive symptoms).
Mindful Attention Awareness Scale | 4 weeks
  Measures mindfulness; mean of 15 items (ranges from 1 to 6, with higher scores indicating greater levels of mindfulness)
Schwartz Outcome Scale | 4 weeks
  Measures general well-being; sum of 10 items (ranges from 0 to 60, with higher scores indicating greater well-being)
Toronto Mindfulness Scale-Decentering Subscale | 1 hour
  Measures decentering; sum of 7 items (higher scores indicate greater levels of decentering)
Opioid Compliance Checklist | 4 weeks
  Measure misuse of opioid medications (scores range from 0 to 12, with higher scoring indicating greater misuse)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided